CLINICAL TRIAL: NCT00742222
Title: Electronic Xoft Intersociety Brachytherapy Trial
Brief Title: Electronic Xoft Intersociety Brachytherapy Trial: Electronic Brachytherapy (EBT) For Treatment of Early Stage Breast Cancer
Acronym: EXIBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR-0186
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer; Carcinoma; Lumpectomy; Ductal Carcinoma in Situ
Keywords: Electronic brachytherapy registry; Multi-society registry; Breast cancer registry
MeSH Terms: conditions — Breast Neoplasms; Carcinoma; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm, treatment with FDA cleared technology (Other): Patients who have early stage breast cancer, and are candidate for intracavitary accelerated partial breast irradiation may be considered for this study.
  Interventions: Radiation: Electronic Brachytherapy; Radiation: Intracavitary accelerated partial breast irradiation

INTERVENTIONS:
Radiation: Electronic Brachytherapy — 34 Gy administered over 10 fractions, twice a day times five days. The radiation therapy treatment will be complete upon the 5th day.
  Other Names: Radiation therapy; APBI; Intracavitary APBI; Accelerated partial breast irradiation; Xoft procedure; Partial breast irradiation; Partial breast radiation therapy; Balloon brachytherapy; Electronic source radiation therapy
Radiation: Intracavitary accelerated partial breast irradiation — 3.4 Gy BID x 5 days
  Other Names: Xoft Axxent system; electronic brachytherapy

SUMMARY:
PRINCIPAL INVESTIGATORS

* Rakesh Patel, MD- Radiation Oncologist
* Peter Beitsch, MD- Breast Surgeon

REGISTRY DESIGN

* Multicenter, non-randomized, post market registry of intracavitary accelerated partial breast irradiation in appropriately selected patients.

SAMPLE SIZE AND SITES:

* Approximately 400 patients may be enrolled.
* Up to 100 qualified U.S. sites may participate in this registry.

ENDPOINTS:

1. PRIMARY ENDPOINTS

   * Subcutaneous Toxicities - The incidence of signs and symptoms of subcutaneous toxicities will be recorded at the following follow-up visits; at six (6) month, one (1) year, two (2) year, three (3) year, four (4) year, and five (5) year.
   * Skin Toxicities - Specific toxicities that can result from radiation therapy will be recorded at each follow-up visit. The Common Terminology Criteria for Adverse Events will be used and to be recorded at each follow-up visits; at one (1) month, six (6) month, one (1) year, two (2) year, three (3) year, four (4) year, and five (5) year.
   * Cosmetic Outcome - Cosmetic outcome will be recorded at the following follow-up visits; at one (1) month, six (6) month, one (1) year, two (2) year, three (3) year, four (4) year, and five (5) year. Cosmetic outcome will be assessed and graded in two ways:
   * Patient Quality of Life Questionnaire - A Quality of Life Questionnaire (QOL) will be completed at the following visits; at one (1) month, six (6) month, one (1) year, two (2) year, three (3) year, four (4) year, and five (5) year.
2. SECONDARY ENDPOINTS

   * Local-regional Breast Failure - The secondary efficacy endpoint is ipsilateral breast failure at five (5) years.

   This includes:
   * Ipsilateral recurrence within the initially treated volume. (Within the tumor bed)
   * Ipsilateral recurrence of cancer outside of the initially treated volume. (Elsewhere Failure)
   * Axillary nodal recurrence

     * Survival - to be recorded at each follow-up visit
   * Overall Survival
   * Disease Free Survival

     * Device Performance - to be recorded during the balloon applicator placement and during the course of the radiation treatments:
   * Ability to deliver treatment
   * Axxent System / Balloon Applicator performance
3. TREATMENT DEVICE

The device to be used is the electronic brachytherapy system for the treatment of early stage breast cancer with intracavitary accelerated partial breast irradiation. The device manufacturer is Xoft, Incorporated. All Xoft technology cleared by the FDA for the treatment of early stage breast cancer can be used in this post market data collection registry.

OVERSIGHT COMMITTEE

Representatives from American Brachytherapy Society (ABS), American Society of Breast Surgeons (ASBS), and American College of Radiation Oncology (ACRO)will oversee study management.

ELIGIBILITY:
Inclusion Criteria:

* Patient 50 years of age or older
* Estrogen receptor positive
* Tumor size ≤ 3cm
* Tumor histology: invasive carcinoma or DCIS
* Patient is node negative
* Patient has negative surgical margins (NSABP definition, no tumor on ink) after final surgery
* Life expectancy > 5 years

Exclusion Criteria:

* Pregnancy or breast-feeding. (If appropriate, patient must use birth control during the registry.) The need for a pregnancy test is based on the physician's standard practice and will be performed according to the physician's standard of care.
* Collagen Vascular Disease
* Scleroderma
* Systemic sclerosis
* Active lupus
* Infiltrating lobular histology
* Previous ipsilateral radiation to the thorax or breast

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The incidence of signs and symptoms of subcutaneous toxicities will be recorded at the following follow-up visits; six month, one year, two year, three year, four year, and five year. | 5 years

SECONDARY OUTCOMES:
Local-regional Breast Failure - Ipsilateral breast failure at five years, Including: Ipsilateral recurrence within the initially treated volume, Ipsilateral recurrence of cancer outside of the initially treated volume, and axillary nodal recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Beitsch, MD, Principal Investigator — Dallas Surgical Group; Rakesh Patel, MD, Principal Investigator — University of Wisconsin Radiation Oncology Department
Locations (8):
- United States (8):
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Beverly Oncology, Montebello, California
  - Florida Radiation Oncology Group, Orange Park, Florida
  - St Elizabeth's and Memorial Cancer Center, Swansea, Illinois
  - Cancer Institute of Cape Girardeau, Cape Girardeau, Missouri
  - AtlantiCare Cancer Care Institute, Galloway, New Jersey
  - Nazha Cancer Center, Northfield, New Jersey
  - Dallas Surgical Group / Northpoint Cancer Center, Dallas, Texas

REFERENCES:
- [Background] Dickler A, Kirk MC, Seif N, Griem K, Dowlatshahi K, Francescatti D, Abrams RA. A dosimetric comparison of MammoSite high-dose-rate brachytherapy and Xoft Axxent electronic brachytherapy. Brachytherapy. 2007 Apr-Jun;6(2):164-8. doi: 10.1016/j.brachy.2007.01.005. PMID 17434111
- [Background] Smitt MC, Kirby R. Dose-volume characteristics of a 50-kV electronic brachytherapy source for intracavitary accelerated partial breast irradiation. Brachytherapy. 2007 Jul-Sep;6(3):207-11. doi: 10.1016/j.brachy.2007.03.002. PMID 17681242